CLINICAL TRIAL: NCT01909349
Title: Rehabiliation-Aftercare for an Optimal Transfer Into Autonomous Daily Life (RENATA) - an eHealth Intervention Study
Brief Title: Web-based Aftercare Intervention for Cardiac Patients
Acronym: RENATA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacobs University Bremen gGmbH (Other)
Collaborators: Maastricht University (Other); Institute of Physical Education and Sports Sciences (Other); Guangdong Provincial People's Hospital (Other); Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Sonia Lippke, Professor of Health Psychology, Jacobs University Bremen gGmbH
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EK-A-SL-022013
Record Dates: First submitted 2013-07-17; First posted 2013-07-26 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: CARDIOVASCULAR DISEASES; HEART DISEASES
Keywords: medical rehabilitation; aftercare; multiple health behavior change; diet; physical activity; computer; international study; ETHNOPSYCHOLOGY; HABIT; HEALTH; eHealth; eLearning
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Motor Activity; Habits | interventions — Professional Autonomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Control Group will gain access to the intervention after the intervention group has finished the program (>8 weeks after signing up)
- Intervention Group I (Experimental): Self-regulation support Behavior sequence: Physical activity, then fruit & vegetable intake
  Interventions: Behavioral: self-regulation

INTERVENTIONS:
Behavioral: self-regulation — Web-based support for behavior change regarding physical activity and fruit & vegetable consumption
  Arms: Intervention Group I

SUMMARY:
Persons undergoing cardiac rehabilitation often have difficulties transferring the learned health behaviors into their daily routine which decreases their health status. Computer-based tailored interventions have been shown to be effective in increasing physical activity as well as fruit and vegetable consumption. The aim of this study is, to support people in transferring these two learned behavior changes and their antecedents into their daily life after cardiac rehabilitation in Germany, the Netherlands and China. The primary goal of the study is to analyze the effectiveness of a rehabilitation aftercare program with regard to the level of physical activity and nutrition.

DETAILED DESCRIPTION:
For cardiac patients, medical rehabilitation after severe medical incidents (e.g., bypass surgery, heart attack, heart failure) is a central part in the recovery process. Health behavior change is an important subject within rehabilitation, and patients have to learn how to improve their eating habits and increase their physical activity. Back home, the adoption, maintenance and transfer into daily life of the behavior change is difficult. Until now it is unclear how such a complex behavior change actually takes place and how it can be supported effectively. On basis of theoretical assumptions (health action process approach, HAPA, Schwarzer, 1992, and compen¬satory carry-over action model, CCAM, Lippke, 2010) multiple behavior change will be observed and supported in an online intervention. To its effects, an intervention will be provided firstly targeting physical activity, secondly nutrition and compared with a waiting-list control group. Furthermore, very little is known about intercultural differences and therefore will be tested with rehabilitation patients with various cultural backgrounds. This all will be archived in the study RENATA.

RENATA is an online based intervention for post-rehabilitative medical care, with the aim to integrate skills and behavior patterns, which were gained during the rehabilitation, into daily life of the participants. The goal is to maintain learning results for a long period of time, improve rehabilitation effects at a sustained basis and support the return to the labor market i.e. to work. The objective of this research project is to increase the self-regulatory abilities of participants to the extent that they are able to be regularly and autonomously physically active and eat healthy, so that they will increase their quality of life and become resilient.

Due to the fact that there is only a limited number of evaluated programs, the present research project has the aim (1) to offer such a program and to test the effectiveness. Moreover, compared on an international level it will be considered (2) if such an aftercare program helps participants equally in different countries with rehabilitation systems varying in intensity. This question will be investigated by comparing Germany, the Netherlands and China. Due to the demographic changes, there are rising numbers of older employees in the labor market who will and should be kept in. Within this context, the last research aim is (3) to examine age effects in detail: Is it possible to determine age-specific differences in the effectiveness of the different interventions?

ELIGIBILITY:
Inclusion Criteria:

* People have Internet access
* People have sufficient knowledge of the Dutch/German language, writing and reading skills
* People have completed cardiac rehabilitation treatment or have suffered from at least one cardiac disease/event in the last 6 months
* People received behavior lifestyle recommendations with regard to physical activity and fruit and vegetable consumption

Exclusion Criteria:

* People who do not want to sign the informed consent
* People with contraindications with regard to physical activity and fruit and vegetable intake
* People without Internet access
* People with insufficient abilities to use computer and Internet
* People with poor cognitive performance/dementia.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in dietary and physical activity behavior (self-report) | Baseline to 8 weeks later
  change scores (mean, residual change) and percentage meeting the recommendations

SECONDARY OUTCOMES:
Body weight | 8 weeks
BMI | 8 weeks
Days of absence from work | 8 weeks
Quality of Life | 8 weeks
Quality of Life | 3 months
Quality of Life | 6 months
Quality of Life | 12 months
Dietary and physical activity behavior (self-report) | 3 months
Dietary and physical activity behavior (self-report) | 6 months
Dietary and physical activity behavior (self-report) | 12 months
Body weight | 3 months
Body weight | 6 months
Body weight | 12 months
Days of absence from work | 3 months
Days of absence from work | 6 months
Days of absence from work | 12 months
BMI | 3 months
BMI | 6 months
BMI | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Lippke, Prof. Dr., Principal Investigator — Jacobs University Bremen
Locations (3):
- China, Hong Kong, Hong Kong, China
- Germany, Bremen, City state Bremen, Germany
- The Netherlands, Maastricht, LK, Netherlands

REFERENCES:
- [Derived] Duan YP, Liang W, Guo L, Wienert J, Si GY, Lippke S. Evaluation of a Web-Based Intervention for Multiple Health Behavior Changes in Patients With Coronary Heart Disease in Home-Based Rehabilitation: Pilot Randomized Controlled Trial. J Med Internet Res. 2018 Nov 19;20(11):e12052. doi: 10.2196/12052. PMID 30455167
- [Derived] Storm V, Reinwand DA, Wienert J, Tan SL, Lippke S. The Mediating Role of Perceived Social Support Between Physical Activity Habit Strength and Depressive Symptoms in People Seeking to Decrease Their Cardiovascular Risk: Cross-Sectional Study. JMIR Ment Health. 2018 Nov 14;5(4):e11124. doi: 10.2196/11124. PMID 30429112
- [Derived] Tan SL, Storm V, Reinwand DA, Wienert J, de Vries H, Lippke S. Understanding the Positive Associations of Sleep, Physical Activity, Fruit and Vegetable Intake as Predictors of Quality of Life and Subjective Health Across Age Groups: A Theory Based, Cross-Sectional Web-Based Study. Front Psychol. 2018 Jun 18;9:977. doi: 10.3389/fpsyg.2018.00977. eCollection 2018. PMID 29967588
- [Derived] Duan YP, Wienert J, Hu C, Si GY, Lippke S. Web-Based Intervention for Physical Activity and Fruit and Vegetable Intake Among Chinese University Students: A Randomized Controlled Trial. J Med Internet Res. 2017 Apr 10;19(4):e106. doi: 10.2196/jmir.7152. PMID 28396306
- [Derived] Kuhlmann T, Reips UD, Wienert J, Lippke S. Using Visual Analogue Scales in eHealth: Non-Response Effects in a Lifestyle Intervention. J Med Internet Res. 2016 Jun 22;18(6):e126. doi: 10.2196/jmir.5271. PMID 27334562
- [Derived] Storm V, Dorenkamper J, Reinwand DA, Wienert J, De Vries H, Lippke S. Effectiveness of a Web-Based Computer-Tailored Multiple-Lifestyle Intervention for People Interested in Reducing their Cardiovascular Risk: A Randomized Controlled Trial. J Med Internet Res. 2016 Apr 11;18(4):e78. doi: 10.2196/jmir.5147. PMID 27068880
- [Derived] Reinwand DA, Crutzen R, Storm V, Wienert J, Kuhlmann T, de Vries H, Lippke S. Generating and predicting high quality action plans to facilitate physical activity and fruit and vegetable consumption: results from an experimental arm of a randomised controlled trial. BMC Public Health. 2016 Apr 12;16:317. doi: 10.1186/s12889-016-2975-3. PMID 27066779
- [Derived] Reinwand D, Kuhlmann T, Wienert J, de Vries H, Lippke S. Designing a theory- and evidence-based tailored eHealth rehabilitation aftercare program in Germany and the Netherlands: study protocol. BMC Public Health. 2013 Nov 19;13:1081. doi: 10.1186/1471-2458-13-1081. PMID 24245493